CLINICAL TRIAL: NCT04699669
Title: A 2-stage, Phase 1/2a Study to Evaluate the Safety, Tolerability, and Preliminary Efficacy of CBL-514 Injection for Reducing Convexity or Fullness of Abdominal Subcutaneous Fat (Phase 1)
Brief Title: A Phase 1 Study to Evaluate the Safety and Tolerability of CBL-514 Injection on Convexity or Fullness of Abdominal Subcutaneous Fat in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Caliway Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: CBL-16001(Phase 1)
Record Dates: First submitted 2020-12-29; First posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: Subcutaneous Fat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Cohort 1: CBL-514 2 mg, 0.5 mg/cm^2 (Other): Individual placebo control. CBL-514 will be administrated with the grid spacing of 4 cm^2
  Interventions: Drug: CBL-514, placebo
- Cohort 2: CBL-514 10 mg, 0.5 mg/cm^2 (Other): Individual placebo control. CBL-514 will be administrated with the grid spacing of 4 cm^2
  Interventions: Drug: CBL-514, placebo
- Cohort 3: CBL-514 20 mg, 0.5 mg/cm^2 (Other): Individual placebo control. CBL-514 will be administrated with the grid spacing of 4 cm^2
  Interventions: Drug: CBL-514, placebo
- Cohort 4: CBL-514 40 mg, 1.0 mg/cm^2 (Other): Individual placebo control. CBL-514 will be administrated with the grid spacing of 4 cm^2
  Interventions: Drug: CBL-514, placebo
- Cohort 5: CBL-514 40 mg, 2 mg/cm^2 (Other): Individual placebo control. CBL-514 will be administrated with the grid spacing of 2 cm^2
  Interventions: Drug: CBL-514, placebo
- Cohort 6: CBL-514 80 mg, 2 mg/cm^2 (Experimental): CBL-514 only. CBL-514 will be administrated with the grid spacing of 2 cm^2
  Interventions: Drug: CBL-514
- Cohort 7: CBL-514 160 mg, 2 mg/cm^2 (Experimental): CBL-514 only. CBL-514 will be administrated with the grid spacing of 2 cm^2
  Interventions: Drug: CBL-514
- Cohort 8: CBL-514 240 mg, 2 mg/cm^2 (Experimental): CBL-514 only. CBL-514 will be administrated with the grid spacing of 2 cm^2
  Interventions: Drug: CBL-514
- Cohort 9: CBL-514 320 mg, 2 mg/cm^2 (Experimental): CBL-514 only. CBL-514 will be administrated with the grid spacing of 2 cm^2
  Interventions: Drug: CBL-514

INTERVENTIONS:
Drug: CBL-514, placebo — One side of the abdominal region will receive CBL-514, while the other will receive placebo with equal volume.
  Which side of the abdominal region to receive CBL-514 or placebo would be randomized.
  No PK samples will be collected in this cohort.
  Arms: Cohort 1: CBL-514 2 mg, 0.5 mg/cm^2; Cohort 2: CBL-514 10 mg, 0.5 mg/cm^2
Drug: CBL-514, placebo — One side of the abdominal region will receive CBL-514, while the other will receive placebo with equal volume.
  Which side of the abdominal region to receive CBL-514 or placebo would be randomized.
  Arms: Cohort 3: CBL-514 20 mg, 0.5 mg/cm^2; Cohort 4: CBL-514 40 mg, 1.0 mg/cm^2; Cohort 5: CBL-514 40 mg, 2 mg/cm^2
Drug: CBL-514 — Both sides of the abdominal region will receive CBL-514.
  Arms: Cohort 6: CBL-514 80 mg, 2 mg/cm^2; Cohort 7: CBL-514 160 mg, 2 mg/cm^2; Cohort 8: CBL-514 240 mg, 2 mg/cm^2; Cohort 9: CBL-514 320 mg, 2 mg/cm^2

SUMMARY:
The Phase 1 component of the study is a double-blind, placebo-controlled, single ascending dose (SAD) design intended to assess the safety, tolerability, and PK of CBL-514. The SAD part will involve 9 proposed dosing cohorts.

DETAILED DESCRIPTION:
The Phase 1 part of the study was a first-in-human, single ascending dose, double-blind, randomized (except Cohorts 6 to 9 [open-label]) study in healthy subjects to evaluate the safety, tolerability and PK of CBL-514, and to determine the dose levels to be used for the Phase 2a part of the study.

ELIGIBILITY:
Inclusion Criteria:

A subject can participate in the study only if all the following criteria are met:

1. Male/female aged 18 years to 64 years old (at Screening), inclusive.
2. Body mass index >18.5 and <35 kg/m2 and body weight ≥50 kg at Screening and Day 1.
3. Has MWC ≥80.0 cm at Screening and Day 1.
4. Subcutaneous fat thickness of at least 3.00 cm (30.0 mm) by pinch method (measured by calibrated caliper) surrounding the navel at Screening and Day 1.
5. Voluntarily signs the Informed Consent Form and, in the opinion of the Investigator or delegate, is physically and mentally capable of participating in the study, and willing to adhere to study procedures.

Exclusion Criteria:

A subject who meets any of the following criteria will not be eligible to enter the study:

1. Female subject of childbearing potential who is not willing to commit to an acceptable contraceptive regimen with her partner from the time of Screening and throughout study participation until 12 weeks after the last study drug dose, or who is currently pregnant or lactating. Male subject who is not willing to commit to an acceptable contraceptive method. Females who have been surgically sterilized (hysterectomy or bilateral oophorectomy) or who are postmenopausal (e.g., defined as at least 50 years with ≥12 months of amenorrhea with a follicle stimulating hormone >40 IU/L) are considered to be of nonchildbearing potential. Subjects who are not of childbearing potential are not required to use contraception.
2. Subject diagnosed with coagulation disorders or is receiving anticoagulant/antiplatelet therapy or medications or dietary supplements, which impede coagulation or platelet aggregation.
3. Subject has diabetes or glycated hemoglobin ≥6.5% (48 mmol/mol) or fasting blood sugar ≥7 mmol/L.
4. Subject has a cardiovascular disease, or shows clinically significant abnormal findings in ECG at Screening.
5. Subject with active or prior history of malignancies (except for successfully treated non-invasive basal cell carcinoma) or being worked-up for a possible malignancy.
6. Subject with a history of human immunodeficiency virus (HIV)-1, hepatitis B, or hepatitis C infections or subjects with active HIV, hepatitis B, or hepatitis C infections at Screening:

   1. Active HIV infection: positive HIV Ag/Ab combo test;
   2. Active hepatitis B virus (HBV) infection: positive HBV surface antigen (HBsAg). Subjects with negative HBsAg but with positive HBV core antibody with or without positive HBV surface antibody will also be excluded. However, subjects with negative HBsAg, negative HBV core antibody, and positive HBV surface antibody may be included.
   3. Active hepatitis C virus (HCV) infection: positive HCV antibody.
7. Subject has abnormal skin or local skin conditions, which in the opinion of Investigator is inappropriate to participate in the study, including but not limited to any of the following:

   1. Skin manifestations of a systemic disease,
   2. Any abnormality of the skin or soft tissues of the abdominal wall in the area to be treated,
   3. Skin or superficial tissue that does not lie flat on its own when the subject is in the supine position,
   4. Sensory loss or dysesthesia in the area to be treated,
   5. Evidence of any cause of enlargement in the abdominal area other than localized subcutaneous fat,
   6. Tattoos on the area to be treated.
8. Subject who has undergone the following procedures:

   1. Previous open or laparoscopic abdominal surgery in the anticipated treatment area,
   2. Cardiac pacemakers or any implantable electrical device,
   3. Metal implants of any type in the area to be treated,
   4. Esthetic procedure to the region to be treated within 6 months before Screening.
9. Subject is on prescription or over-the-counter weight reduction medication or weight reduction programs within 3 months before Screening.
10. Subject is undergoing chronic steroid or immunosuppressive therapy.
11. Requiring continual use of the following therapeutic agents during the study:

    S-mephenytoin, terfenadine, buspirone, fexofenadine, breast cancer resistance protein (BCRP) substrates (such as mitoxantrone, methotrexate, topotecan, nitrofurantoin, dipyridamole, statins, etc.), cytochrome P450 3A4 inhibitor, or non-steroidal anti-inflammatory drugs (NSAIDs). If a subject needs to use the above mentioned therapeutic agents during the study for any reason, these therapeutic agents should not be used at least for 48 hours prior to dosing until 24 hours post-dose or the collection of the last PK sample, whichever is later.
12. Unable to receive topical anesthesia (e.g., history of hypersensitivity to lidocaine).
13. Subjects with known allergies or sensitivities to the study drug and/or excipients.
14. Subjects with inadequate liver function at Screening defined as aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total bilirubin, or gamma-glutamyl transferase >1.5 × ULN. A subject with an elevated liver chemistry test up to 1.5 × ULN at Screening should be evaluated by the Investigator to exclude pre-existing liver disease associated with mild elevation of liver chemistry tests. If the mild elevation is assessed by the Investigator as not clinically significant or related to non-alcoholic fatty liver, the subject may be eligible if the follow-up tests show an unchanged or reducing value from the initial Screening value. A subject with marginally elevated fasting unconjugated serum bilirubin with documented Gilbert's syndrome, and no other cause for the elevated bilirubin on investigation, may be eligible.
15. Subjects with inadequate renal function, defined as abnormal serum creatinine, and urea >1.5 × ULN or estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2.

    Subjects who are currently on dialysis should be excluded. A subject with serum urea between 1 to 1.5 × ULN at Screening, but an eGFR >60mL/min/1.73 m2 and no other renal risk factors, should be re-tested prior to declaring the subject as eligible. The subject may be eligible if the fasting serum creatinine is not rising nor the eGFR falling, the urinary albumin/creatinine ratio remain <3 mg/mmol.
16. Use of other investigational drug or device within 4 weeks prior to Screening.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-27 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to 4 weeks after treatment
  Number of participants experiencing TEAEs and number of individual TEAEs among treatment groups by severity and relationship to investigational product (IP)
Number of participants with clinically significant abnormalities in clinical laboratory values | Up to 2 weeks after treatment
  Clinical laboratory tests include Biochemistry, Hematology, Coagulation and Urinalysis testinjection site reactions.
Number of participants with clinically significant abnormalities in vital signs | Up to 2 weeks after treatment
  Vital signs measurements include temperature, pulse rate, blood pressure, and respiratory rate
Number of participants with clinically significant abnormalities in Electrocardiogram (ECG) | Up to 2 weeks after treatment
  ECG parameters include heart rate, RR interval, PR interval, QT interval, QTc interval, and QRS interval
Number of participants with clinically significant abnormalities in physical examination | Up to 2 weeks after treatment
  Physical examinations include assessment of cardiovascular, respiratory, gastrointestinal, and neurological systems
Number of participants with injection site reactions | Up to 2 weeks after treatment
  Injection site reactions include but not limited to redness, swelling, bruising, tenderness, itching, pain, warmth, discoloration and hardness

SECONDARY OUTCOMES:
Assess maximum concentration of CBL-514 in plasma (Cmax) | Up to 24 hours after treatment
  To evaluate maximum concentration of CBL-514 in plasma (Cmax) after single dose injection.
Assess time to Cmax of CBL-514 in plasma (tmax) | Up to 24 hours after treatment
  To evaluate time to Cmax of CBL-514 in plasma (tmax) after single dose injection.
Assess area under the concentration-time curve of CBL-514 in plasma (AUC) | Up to 24 hours after treatment
  To evaluate area under the concentration-time curve of CBL-514 in plasma (AUC) after single dose injection.
Assess terminal rate constant and half-life of CBL-514 in plasma (λz and t1/2) | Up to 24 hours after treatment
  To evaluate terminal rate constant and half-life of CBL-514 in plasma (λz and t1/2) after single dose injection.
Assess apparent clearance and volume of distribution of CBL-514 in plasma (CL/F and Vz/F). | Up to 24 hours after treatment
  To evaluate apparent clearance and volume of distribution of CBL-514 in plasma (CL/F and Vz/F) after single dose injection.

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: No